CLINICAL TRIAL: NCT05602246
Title: Study Comparing Transobturator Cystocele vs. Anterior Vaginal RepairS
Acronym: STARS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Zdenek Rusavy, assoc. prof. MD PhD, Charles University, Czech Republic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STARS
Record Dates: First submitted 2022-10-23; First posted 2022-11-02 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Pelvic Organ Prolapse; Cystocele; Cystocele and Incomplete Uterovaginal Prolapse
Keywords: Pelvic organ prolapse; Quality of life; TOCR; Anterior vaginal wall repair; Transobturator cystocele repair
MeSH Terms: conditions — Pelvic Organ Prolapse; Cystocele

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transobturator cystocele repair (TOCR) (Experimental): The technique of TOCR was published previously including a video [Kalis et al. Trans-obturator cystocele repair (TOCR) of level 2 paravaginal defect. Int Urogynecol J. 2020, 31(11):2435-38. doi:10.1007/s00192-020-04337-x].
  The anterior vaginal wall is incised in the midline and the pubocervical fascia is dissected to open the paravaginal space towards the ATFP and the fascia of the obturator internus muscle. 3-4 continuous non-locking stitches of non-absorbable suture 1-0 Ti-Cron™ braided polyester are taken into the pubocervical fascia and threaded using Shirodkar needles through skin incisions in genitofemoral sulci passing through the full thickness of the obturator membrane, obturator internus muscle. After closure of the vaginal skin incision, both ends of the Ti-Cron™ sutures are tied ensuring the obliteration of the paravaginal defect.
  Indometacin rectal suppository 100 mg is inserted transrectally for early postoperative pain management.
  Interventions: Procedure: Transobturator cystocele repair
- standard anterior colporrhaphy (anterior repair - AR) (Active Comparator): The anterior vaginal wall is incised in the midline from the level of the bladder neck up to vaginal apex or anterior vaginal fornix. The bladder is sharply dissected from the vaginal wall with pubocervical fascia attached to the bladder wall. The fascia is approximated in the midline with several simple interrupted 0 polyglactin 910 sutures or equivalent. The surplus of distended vaginal epithelium is trimmed. The vaginal incision is closed using a continuous non-locking polyglactin 910 2-0 suture or equivalent. Indometacin rectal suppository 100 mg is inserted transrectally for early postoperative pain management.
  Interventions: Procedure: Anterior colporrhaphy

INTERVENTIONS:
Procedure: Transobturator cystocele repair — Novel transvaginal surgical reconstruction of anterior compartment pelvic organ prolapse.
  Other Names: TOCR
  Arms: Transobturator cystocele repair (TOCR)
Procedure: Anterior colporrhaphy — The traditional transvaginal surgery for cystocele treatment used as a comparator in the study
  Other Names: Anterior repair
  Arms: standard anterior colporrhaphy (anterior repair - AR)

SUMMARY:
Surgical correction of the prolapse in the anterior compartment remains one of the major challenges in urogynecology. Paravaginal defect in level II of vaginal fixation results in the majority of cystoceles. Clinically, these defects are often combined and/or may be bilateral. Hence, careful assessment and individualized planning of the surgical procedure is essential to optimize cystocele repair outcome. Several surgical techniques and approaches have been used for cystocele repair. After the ban on transvaginal meshes, the interest in native tissue repair has risen. Paravaginal defect repair is an effective surgery for paravaginal defect reconstruction. There is a current trend to utilize transvaginal surgery instead of more invasive transabdominal surgery. A novel method of transvaginal paravaginal defect repair - TOCR (transobturator cystocele repair) was suggested. The principle objective of the present trial is to compare its efficacy and safety to preexisting method of native tissue cystocele repair.

DETAILED DESCRIPTION:
Pelvic organ prolapse (POP) has a negative impact on the quality of life of affected women and anterior compartment defects remain the most challenging to repair. It was reported that a women has almost a 1 in 5 risk of needing any kind of POP surgery in her lifetime, with anterior wall repair accounting for 40.6% of all of these. Depending on the structures affected, cystocele can be secondary to defects at: A) Level I vaginal support, provided by the uterosacral and cardinal ligaments or B) Level II vaginal support, mainly provided by the pubocervical fascia. Level II defects can be midline or lateral (paravaginal) depending on whether the fascia is weak at the midline or detached from its lateral attachment to the arcus tendineus fasciae pelvis (ATFP). Clinically, these defects are often combined and/or may be bilateral. Hence, careful assessment and individualized planning of the surgical procedure is essential to optimize cystocele repair outcome.

Several surgical techniques and approaches have been used for cystocele repair. These involve native tissue and the use of mesh implanted transvaginally and / or transabdominally.The mainstay for the vaginal repair of a level I defects is to anchor the uterine cervix or vaginal vault to the sacrospinous or the anterior longitudinal ligaments. However, proper restoration of a level II defect is more complex. Although, a classical anterior colporrhaphy might be suitable to correct an isolated midline weakness in the endopelvic fascia, it is suboptimal, on its own, for the repair an associated lateral defect, which is a common association. Indeed, De Lancey reported that paravaginal defects (PVDs) were diagnosed in 89% of women undergoing surgery for cystocele and stress urinary incontinence.

Although a variety of techniques for paravaginal defect repair (PVDR) have been suggested, several of these are now not feasible in many countries following the FDA's ban on transvaginal mesh manufacture, sale and distribution. Therefore, currently there are attempts to utilize minimally invasive approaches and modern devices in PVDR native tissue repair. Applying this principle, e.g. Capio Suture Capturing Device (Boston Scientific) has been proposed to re-attach the vagina to the ATFP using two to four non-absorbable sutures. However, based on anatomical observation, the ATFP is thin its superior part and thicker inferiorly. This is an issue that might affect the reliability of identifying and ensuring a secure anchorage to the ATFP when solely using a transvaginal route. Recently a novel. Technique of PVDR, called transobturator cystocele repair has been published. However, as the technique was described recently, no follow-up data have been reported to support its practice.

The aim of this randomized controlled trial (RCT) is to compare the novel TOCR and standard anterior colporrhaphy (AR) regarding their safety, efficacy and quality-of-life improvement in a one-year follow-up.

ELIGIBILITY:
Inclusion Criteria:

* (at least) 2nd stage prolapse of the anterior compartment (Ba ≥ -1)
* Age ≥ 50 years
* Symptom bulge
* Ability to speak Czech or English

Exclusion Criteria:

* Malignancy

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 592 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Anatomic failure | 1 year
  Anterior compartment pelvic organ prolapse stage ≥ 2( i.e. pelvic organ prolpase quantification (POPQ) point Ba, or C of > -1)

SECONDARY OUTCOMES:
Composite surgery failure | 1 year
  Composite measure requiring at least one from the following: 1. anatomic failure (Pelvic Organ Prolapse Quantification point Ba, Bp, or C of > 0), 2. subjective failure (presence of bothersome vaginal bulge symptoms), or 3. pessary or surgical retreatment for pelvic organ prolapse
2-year composite surgery failure | 2 years
  Composite measure requiring at least one from the following: 1. anatomic failure (Pelvic Organ Prolapse Quantification point Ba, Bp, or C of > 0), 2. subjective failure (presence of bothersome vaginal bulge symptoms), or 3. pessary or surgical retreatment for pelvic organ prolapse
2-year anatomic failure | 2 years
  Anterior compartment pelvic organ prolapse stage ≥ 2( i.e. POPQ point Ba, or C of > -1)
Complication rate | 1 year
  Number of complications Dindo-Clavien Grade > 2
Pain after the surgery | Postoperative day 14
  visual analog scale (VAS) ≥ 3 (range 0-10, higher is worse)
Subjective perception of improvement | 1 year
  Patient global impression of improvement (PGI-I) ≤ 2 (range 1-7, higher is worse)
2-year subjective perception of improvement | 2 years
  PGI-I ≤ 2 (range 1-7, higher is worse)
Patient satisfaction | 1 year
  Subjectively assessed by the patient on a scale 0 - 100%. Satisfaction with the surgery ≥ 80 %.
De novo stress urinary incontinence (SUI) | 1 year
  Any new stress leaks of urine reported by the patient ≥ once a week, or treatment
De novo overactive bladder (OAB) | 1 year
  de novo OAB ≥ once a week, or treatment
Change in quality of life - urinary incontience | 1 year
  assessed by Urinary Distress Inventory (UDI-6) score, range 0-100, higher is worse
Change in quality of life - prolapse bother | 1 year
  assessed by Pelvic Organ Prolapse Distress Inventory (POPDI-6) score, range 0-100, higher is worse
Change in quality of life - anorectal problems | 1 year
  assessed by Colorectal-Anal Distress Inventory (CRADI-8) score,range 0-100, higher is worse.
Change in quality of sexual life | 1 year
  assessed by Pelvic Organ Prolapse/Incontinence Sexual Questionnaire, IUGA-Revised (PISQ-IR) single summary score in sexually active women (higher is better)
Change in severity of urinary incontinence | 1 year
  assessed by International Consultation of Incontinence Questionnaire - Short Form (ICIQ-UI SF) score (0-21, higher is worse)

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Kalis, prof. MD PhD, Study Chair — Faculty of Medicine in Plzen, Charles University; Khaled MK Ismail, MBBCh, MSc, MD, PhD, FRCOG, Study Director — Faculty of Medicine in Plzen, Charles University; Zdenek Rusavy, assoc. prof. MD PhD, Principal Investigator — Faculty of Medicine in Plzen, Charles University
Locations (8):
- Czechia (6):
  - Faculty of Medicine in Hradec Kralove, Charles University, Hradec Králové
  - Medical Faculty, Ostrava University, Ostrava-Poruba
  - Hospital Pardubice Region, Inc., Pardubice
  - Faculty of Medicine in Pilsen, Charles University, Pilsen
  - Hospital na Bulovce, 1st Medical Faculty, Charles University, Prague
  - Tomas Bata Regional Hospital in Zlin, Zlín
- Slovakia (2):
  - Košice Medical University, Košice
  - Trenčianska univerzita Alexandra Dubčeka, Trenčín

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lowenstein E, Ottesen B, Gimbel H. Incidence and lifetime risk of pelvic organ prolapse surgery in Denmark from 1977 to 2009. Int Urogynecol J. 2015 Jan;26(1):49-55. doi: 10.1007/s00192-014-2413-y. Epub 2014 May 20. PMID 24842118
- [Background] Otcenasek M, Gauruder-Burmester A, Haak LA, Grill R, Popken G, Baca V. Paravaginal defect: A new classification of fascial and muscle tears in the paravaginal region. Clin Anat. 2016 May;29(4):524-9. doi: 10.1002/ca.22694. Epub 2016 Feb 14. PMID 26800142
- [Background] Arenholt LTS, Pedersen BG, Glavind K, Glavind-Kristensen M, DeLancey JOL. Paravaginal defect: anatomy, clinical findings, and imaging. Int Urogynecol J. 2017 May;28(5):661-673. doi: 10.1007/s00192-016-3096-3. Epub 2016 Sep 17. PMID 27640064
- [Background] Arenholt LTS, Pedersen BG, Glavind K, Greisen S, Bek KM, Glavind-Kristensen M. Prospective evaluation of paravaginal defect repair with and without apical suspension: a 6-month postoperative follow-up with MRI, clinical examination, and questionnaires. Int Urogynecol J. 2019 Oct;30(10):1725-1733. doi: 10.1007/s00192-018-3807-z. Epub 2018 Dec 1. PMID 30506182
- [Background] de Tayrac R, Boileau L, Fara JF, Monneins F, Raini C, Costa P. Bilateral anterior sacrospinous ligament suspension associated with a paravaginal repair with mesh: short-term clinical results of a pilot study. Int Urogynecol J. 2010 Mar;21(3):293-8. doi: 10.1007/s00192-009-1036-1. PMID 19924370
- [Background] Ward RM, Sung VW, Clemons JL, Myers DL. Vaginal paravaginal repair with an AlloDerm graft: Long-term outcomes. Am J Obstet Gynecol. 2007 Dec;197(6):670.e1-5. doi: 10.1016/j.ajog.2007.08.067. PMID 18060976
- [Background] Chinthakanan O, Miklos JR, Moore RD. Laparoscopic Paravaginal Defect Repair: Surgical Technique and a Literature Review. Surg Technol Int. 2015 Nov;27:173-83. PMID 26680393
- [Background] Delancey JO. Fascial and muscular abnormalities in women with urethral hypermobility and anterior vaginal wall prolapse. Am J Obstet Gynecol. 2002 Jul;187(1):93-8. doi: 10.1067/mob.2002.125733. PMID 12114894
- [Background] Holt E. US FDA rules manufacturers to stop selling mesh devices. Lancet. 2019 Apr 27;393(10182):1686. doi: 10.1016/S0140-6736(19)30938-9. No abstract available. PMID 31034366
- [Background] Leffler KS, Thompson JR, Cundiff GW, Buller JL, Burrows LJ, Schon Ybarra MA. Attachment of the rectovaginal septum to the pelvic sidewall. Am J Obstet Gynecol. 2001 Jul;185(1):41-3. doi: 10.1067/mob.2001.116366. PMID 11483901
- [Background] Kalis V, Kovarova V, Rusavy Z, Ismail KM. Trans-obturator cystocele repair of level 2 paravaginal defect. Int Urogynecol J. 2020 Nov;31(11):2435-2438. doi: 10.1007/s00192-020-04337-x. Epub 2020 Jun 3. PMID 32494957
- [Background] Jelovsek JE, Gantz MG, Lukacz E, Sridhar A, Zyczynski H, Harvie HS, Dunivan G, Schaffer J, Sung V, Varner RE, Mazloomdoost D, Barber MD; Eunice Kennedy Shriver National Institute of Child Health and Human Development Pelvic Floor Disorders Network. Success and failure are dynamic, recurrent event states after surgical treatment for pelvic organ prolapse. Am J Obstet Gynecol. 2021 Apr;224(4):362.e1-362.e11. doi: 10.1016/j.ajog.2020.10.009. Epub 2020 Oct 8. PMID 33039390
- [Result] Delacroix C, Allegre L, Chatziioannidou K, Gerard A, Fatton B, de Tayrac R. Anterior bilateral sacrospinous ligament fixation with concomitant anterior native tissue repair: a pilot study. Int Urogynecol J. 2022 Dec;33(12):3519-3527. doi: 10.1007/s00192-022-05092-x. Epub 2022 Feb 28. PMID 35226145